CLINICAL TRIAL: NCT05698329
Title: A Phase 1 Study of the Safety, Pharmacokinetics, and Exploratory Efficacy of Periocular Administration of AIV007 in Subjects with Macular Edema Secondary to Neovascular Age-Related Macular Degeneration (nAMD) or Diabetic Macular Edema (DME)
Brief Title: Effect of AIV007 by Periocular Administration in Subjects with Macular Edema Secondary to Neovascular Age-related Macular Degeneration (nAMD) and Diabetic Macular Edema (DME)
Acronym: DME
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AiViva BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AIV007-E02
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-12

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema; Macular Edema
Keywords: Anti-VEGF inhibitor; nAMD; Macular edema; DME; periocular; drug depot
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Intervention Model Description: Route of administration is by delivering single injection of AIV007 in the periocular tissue anatomically juxtasclearal where by the drug depot forms and delivers active agent over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- AIV007 low dose (Experimental): Periocular injection, low dose
  Interventions: Drug: AIV007
- AIV007 intermediate dose 1 (Experimental): Periocular injection, intermediate dose 1
  Interventions: Drug: AIV007
- AIV007 intermediate dose 2 (Experimental): Periocular injection, intermediate dose 2
  Interventions: Drug: AIV007
- AIV007 intermediate dose 3 (Experimental): Periocular injection, intermediate dose 3
  Interventions: Drug: AIV007
- AIV007 intermediate dose 4 (Experimental): Periocular injection, intermediate dose 4
  Interventions: Drug: AIV007
- AIV007 High dose (Experimental): Periocular injection, high dose
  Interventions: Drug: AIV007

INTERVENTIONS:
Drug: AIV007 — Periocular injection

SUMMARY:
To determine safety, pharmacokinetics, and duration of effect of periocularly administered AIV007 gel suspension in subjects with neovascular age-related macular degeneration (nAMD) or diabetic macular edema (DME).

DETAILED DESCRIPTION:
AIV007 is a multiple kinase inhibitor of vascular endothelial growth factor receptors (VEGFR 1, -2 & -3); fibroblast growth factor receptors (FGFR-1, -2, -3 & -4); and platelet-derived growth factor receptors (PDGFR-α & β)1. Lenvatinib is the active pharmaceutical ingredient in AIV007 formulation that is FDA-approved for oral administration for patients with advanced renal cell carcinoma (RCC), differentiated thyroid cancer (DTC), unresectable hepatocellular carcinoma (HCC), and advanced endometrial carcinoma (Lenvima USPI 2021; NDA 206947).

AiViva BioPharma, Inc. (AiViva) has developed a novel, thermoresponsive gel suspension of AIV007 for periocular administration to form a durable depot. This monotherapy is in development for the treatment of retinal and choroidal vascular disease (i.e., neovascular age-related macular degeneration (nAMD) & diabetic macular edema (DME)). For preclinical and clinical (AIV007-E02) studies using periocular administration, AIV007 is injected outside the eyeball and the depot forms a soft mass, referred to as posterior juxtascleral depot (PJD) placement.

ELIGIBILITY:
Inclusion Criteria:

General inclusion Criteria:

1. Male or female subjects aged 21-90 years (inclusive) at screening
2. BCVA in the study eye at screening and baseline/Day 1: ETDRS letter score ≤ 75 and ≥ 24 (20/32 to 20/330 Snellen equivalent)
3. Subject must have received treatment within the 24 months before screening with intravitreal (IVT) injections of an anti-VEGF agent with the last anti-VEGF injection in the study eye being at least 6 weeks (42 days) before baseline/Day 1.
4. Subject has documentation of anti-VEGF responsiveness
5. Subject must provide written informed consent before any study-related procedures are performed
6. Clear ocular media and adequate pupil dilation in both eyes to permit good-quality photographic imaging

nAMD subject

1. The active CNV is confirmed by FA (evidence of leakage)
2. Residual intraretinal or subretinal fluid based on SD-OCT
3. CST ≥ 300 µm as assessed by SD-OCT
4. Total lesion size < 10 disc areas (25.4 mm2)
5. Absence of geographic atrophy within 200 µm of the fovea
6. If subretinal hemorrhage is present, it must be < 50% of the total CNV lesion and/or not involve the fovea
7. If fibrosis is present, it must be <50% of the total lesion area

DME subject

1. Diagnosis of diabetes mellitus (Type 1 or Type 2)
2. Subject has clinically significant DME with central involvement (CST≥300 μm by OCT)
3. The decrease in vision in the study eye was determined by the investigator to be primarily the result of DME

Exclusion Criteria:

1. Previous treatment for nAMD or DME in the study eye other than standard-of-care anti-VEGF IVT injection, e.g., cell therapy, brachytherapy, gene therapy
2. Uncontrolled IOP, defined as an IOP > 25 mmHg
3. Poorly controlled diabetes mellitus defined as hemoglobin A1c (HbA1c) >10% at screening visit
4. The spherical equivalent for refractive error in the study eye of worse than 8.0 diopters of myopia (before cataract or refractive surgery) per the current prescription
5. Any history of active bacterial, viral, fungal, or parasitic ocular or periocular infection, or intraocular inflammation in either eye within the 30 days before the screening Visit
6. History of vitreous hemorrhage within 3 months before screening in the study eye
7. Uncontrolled systemic disease or any other condition or therapy that would make the participant unsuitable for the study
8. Participation in any investigational study within 60 days before the screening visit, or planned use of an investigational product or device during the study; any exposure to a prior investigational drug product must be fully washed out (at least 5 half-lives)
9. History of allergy or hypersensitivity to constituents of the study treatment formulation, topical iodine, ocular antimicrobial solutions, or clinically relevant hypersensitivity to fluorescein

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Approximately 168 days
  Incidence of adverse events and serious adverse events

SECONDARY OUTCOMES:
Mean change from baseline in best-corrected visual acuity (BCVA) | Approximately 168 days
  Number of Early Treatment Diabetic Retinopathy Study (ETDRS) letters
Mean change from baseline in central subfield thickness as measured by spectral domain optical coherence tomography (SD-OCT) | Approximately 168 days
  SD-OCT read by a central reading center
Mean time to rescue medication | Approximately 168 days
  number of days to receive rescue medication

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Retina-Vitreous Associates, Beverly Hills, California
  - Orange County Retina, Santa Ana, California
  - Verum Research, Eugene, Oregon
  - Valley Retina Institute, McAllen, Texas
  - Texas Retina Associates, Plano, Texas
  - Medical Center Ophthalmology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No